CLINICAL TRIAL: NCT04583033
Title: Lifestyle Stressors of Hippocampus and Alzheimer's Disease (AD) Related Brain Regions: Potential for Intervention
Brief Title: Sleep Well for Healthy Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Florida Department of Health (Other Government)
Responsible Party: Principal Investigator, Noam Alperin, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20201031
Record Dates: First submitted 2020-10-06; First posted 2020-10-12 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Poor Quality Sleep
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy (CBT) Group (Experimental): Participants will receive CBT intervention bi-weekly for total of six (6) sessions.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Control Group (No Intervention): Participants will not receive any intervention as part of the study.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — Treatment components include stimulus control, sleep restriction therapy, relaxation, and cognitive therapy. Each session will last approximately one hour and will be provided on line.
  Arms: Cognitive Behavioral Therapy (CBT) Group

SUMMARY:
The purpose of this study is to slow down the aging of the participant's brain by improving sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking healthy subjects age 55 years and older capable and willing to consent to participate in the study. In addition, subject should be cognitively normal and have well documented sleep issues that results with poor sleep quality based on self-reported assessment.

Exclusion Criteria:

* pregnant women
* cognitively impaired subjects not able to provide consent
* prisoners
* Subjects 55 years of age and older that meet criteria for mild cognitive impairment.
* Subjects with any neurological disorder.
* Any other condition that in the opinion of the investigator may affect the participation in this study

Ages: 55 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Rate of brain tissue volume loss in specific brain regions | Year 2
  As evaluated from the Magnetic Resonance Imaging (MRI) Brain scan

SECONDARY OUTCOMES:
Cognitive Performance | Year 2
  Cognitive performance will be assessed using a Memory test which has a composite score ranging from 80 to 120 % with a higher score indicating better performance and a midrange at 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Noam Alperin, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No